CLINICAL TRIAL: NCT04728347
Title: A Phase 2a, Open Label Extension Study to Assess the Safety and Long-Term Immunogenicity of ARCT-021
Brief Title: Open Label Extension Study to Assess the Safety and Long-Term Immunogenicity of ARCT-021
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A decision was made to terminate the study for operational/business reasons. This study was not terminated for reasons of safety or immunogenicity.
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARCT-021-02
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARCT-021 (Experimental): Participants will receive a single dose of ARCT-021 on Day 1
  Interventions: Biological: ARCT-021
- Long-term follow up from ARCT-021-01 (No Intervention): Participants will not receive intervention but will be followed for safety.

INTERVENTIONS:
Biological: ARCT-021 — ARCT-021 single dose
  Arms: ARCT-021

SUMMARY:
This is an open-label study enrolling healthy adults that participated in Study ARCT-021-01 (the Parent Study). Participants will receive either a single injection of ARCT-021 or no injection and be followed for up to 365 days.

DETAILED DESCRIPTION:
This is a phase 2a, open-label study enrolling up to 106 healthy adults that participated in Study ARCT-021-01 (the Parent Study). Participants will enter this study approximately 3 months after their final study visit in the Parent Study. Participants that received placebo in the Parent Study or who are seronegative for SARS-CoV-2 neutralizing antibodies at screening will receive a single dose of ARCT-021 and will be followed for 365 days. Participants that received two injections of ARCT-021 in the Parent Study will not receive any further injections of ARCT-021 and will be followed for 281 days.

ELIGIBILITY:
Inclusion Criteria:

Individuals who:

1. are able to give consent
2. must have completed Study ARCT-021-01
3. agree to comply with all study visits and procedures

   Only for subjects that will receive ARCT-021 in this study:
4. are healthy and medically stable
5. are not planning to donate blood or plasma until 28 days after the last dose of ARCT-021.
6. are willing to refrain from strenuous exercise/activity and alcohol for at least 72 hours prior to study visits and until 28 days after the last dose of ARCT-021.
7. are willing to adhere to contraception requirements if sexually active and/or are of child-bearing potential

Exclusion Criteria:

Individuals who:

1. are unable to comply with the study visits or procedures in Study ARCT-021-01
2. received placebo in the Parent Study and who are not willing to receive ARCT-021 in this study.

   Only for subjects that will receive ARCT-021 in this study:
3. have or will receive any of the SARS CoV-2 or another experimental coronavirus during this study.
4. have a diagnosis of new clinically significant abnormalities including but not limited to

   * Respiratory disease requiring daily medications or oxygen currently or any treatment of respiratory disease exacerbations
   * Significant heart conditions
   * Significant neurological conditions
   * Significant blood disorders
   * Newly diagnosed autoimmune disease
   * Major surgery
5. have abnormal screening laboratory results
6. have uncontrolled diabetes
7. use of any prescription or over-the-counter medications within 7 days prior to vaccination
8. have received immunoglobulins and/or any blood or blood products
9. have a bleeding disorder
10. have uncontrolled blood pressure
11. have been treated with another investigational drug, biological agent, or device since completion of the Parent Study
12. have received or plan to receive:

    * A licensed, live vaccine within 4 weeks before or after study vaccination, or
    * A licensed, inactivated vaccine within 2 weeks before or after study vaccination
13. have traveled outside of Singapore within 30 days before the vaccination or plans to travel outside of Singapore within 60 days after vaccination.
14. other restrictions may apply

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SingHealth Investigational Medicine Unit (IMU), Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1a: Participants who participated in Study ARCT-021-01 (the Parent Study [NCT04480957]) and were without detectable neutralizing antibody responses at baseline received a single-dose primary injection of ARCT-021 on Day 1.
- Cohort 1b: Participants who participated in Study ARCT-021-01 (the Parent Study [NCT04480957]) and were without detectable neutralizing antibody responses at baseline received a single-dose booster injection of ARCT-021 on Day 1.
- Cohort 2 Younger Adults: Participants aged 21 to 55 years old who participated in Study ARCT-021-01 (the Parent Study [NCT04480957]) and were vaccinated with ARCT-021 who did not receive subsequent vaccination with ARCT-021 in this study.
- Cohort 2: Older Adults: Participants aged 56 to 80 years old who participated in Study ARCT-021-01 (the Parent Study [NCT04480957]) and were vaccinated with ARCT-021 who did not receive subsequent vaccination with ARCT-021 in this study.
Period: Overall Study
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2 Younger Adults | Cohort 2: Older Adults
Started | 12 | 12 | 25 | 16
Received Study Drug in This Study | 12 | 12 | 0 | 0
Completed | 12 | 12 | 24 | 16
Not Completed | 0 | 0 | 1 | 0
Not completed — Sponsor decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data presented for all enrolled participants. As pre-specified, baseline characteristics are presented per sub-cohort (younger and older adults) for Cohort 2.
Groups:
- Cohort 2: Younger Adults: Participants aged 21 to 55 years old who participated in Study ARCT-021-01 (the Parent Study [NCT04480957]) and were vaccinated with ARCT-021 who did not receive subsequent vaccination with ARCT-021 in this study.
- Total: Total of all reporting groups
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2: Younger Adults | Cohort 2: Older Adults | Total
Number analyzed (Participants) | 12 | 12 | 25 | 16 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (14.99) | 48.3 (16.17) | 39.7 (8.34) | 63.7 (4.13) | 48.2 (14.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 9 | 4 | 18
  Male | 9 | 10 | 16 | 12 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 25 | 16 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 12 | 11 | 22 | 16 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 1 | 1 | 0 | 2
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Events
Description: Solicited local adverse events were defined as pain, tenderness, erythema, or swelling at the injection site. Solicited systemic adverse events were defined as fever, fatigue, headache, chills, nausea, vomiting, diarrhoea, myalgia, and arthralgia. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to Day 7 (7 days after vaccine administration)
Population: Safety population for Cohort 1a, which included all participants who received Study vaccine in ARCT-021-02 only, and in the Longitudinal Safety population for Cohort 1b, which included all participants who received Study vaccine in ARCT- 021-01 and ARCT-021-02. As pre-specified, data is reported for Cohort 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a | Cohort 1b
Number analyzed (Participants) | 12 | 12
Participants
  Solicited Local | 11 | 10
  Solicited Systemic | 11 | 8

2. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Unsolicited adverse events were defined as any spontaneously occurring adverse event (serious and non-serious). A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to Day 29 (28 days after vaccine administration)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a | Cohort 1b
Number analyzed (Participants) | 12 | 12
Participants | 3 | 2

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), Unsolicited Adverse Events Associated With New Onset of Chronic Disease (NOCD) or Medically Attended Adverse Events (MAAEs)
Description: SAEs were defined as any event that resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, a congenital anomaly or birth defect, or was an important medical event. A NOCD was defined as a MAAE that led to the new diagnosis of a chronic medical condition that was not present or suspected prior to enrollment. A MAAE was an adverse event that led to an unscheduled visit (including a telemedicine visit) to a healthcare practitioner. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to a maximum of approximately 12 months
Population: Safety population for Cohort 1a, which included all participants who received Study vaccine in ARCT-021-02 only, and in the Longitudinal Safety population for Cohorts 1b and Cohort 2, which included all participants who received Study vaccine in ARCT- 021-01 and ARCT-021-02 (Cohort 1b) or ARCT-021-01 only (Cohort 2).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2: Younger Adults | Cohort 2: Older Adults
Number analyzed (Participants) | 12 | 12 | 25 | 16
Participants
  SAEs | 0 | 1 | 0 | 0
  Unsolicited Adverse Events Associated with NOCD | 0 | 1 | 0 | 0
  MAAEs | 2 | 5 | 3 | 0

4. Secondary Outcome: Geometric Mean Titer (GMT) of Serum Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Neutralizing Antibodies
Time Frame: Cohorts 1a and 1b: Days 1, 29, 57, Cohort 2: Day 29
Population: Immunogenicity population, which included all participants who received Study vaccine in either ARCT-021-01 or ARCT-021-02 who had evaluable immunogenicity data following first vaccine administration. Overall number of participants analyzed' = participants evaluable for endpoint. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2: Younger Adults | Cohort 2: Older Adults
Number analyzed (Participants) | 11 | 11 | 19 | 3
Titer
  Day 1: number analyzed (Participants) | 11 | 11 | 0 | 0
  Day 1 | 5.0 [5.00 to 5.00] | 7.3 [3.14 to 16.99] |  |
  Day 29 | 6.1 [4.46 to 8.41] | 38.6 [12.10 to 123.12] | 9.7 [4.28 to 21.75] | 5.0 [5.00 to 5.00]
  Day 57: number analyzed (Participants) | 10 | 10 | 0 | 0
  Day 57 | 5.7 [4.28 to 7.45] | 23.5 [7.65 to 71.98] |  |

5. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in SARS-CoV-2 Neutralizing Antibody Titers
Time Frame: Cohort 1a: Days 29, 57, Cohort 1b: Days 1, 29, 57, and Cohort 2: Day 29
Population: Immunogenicity population, which included all participants who received Study vaccine in either ARCT-021-01 or ARCT-021-02 and had evaluable immunogenicity data following first vaccine administration. Overall number of participants analyzed' = participants evaluable for endpoint. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2: Younger Adults | Cohort 2: Older Adults
Number analyzed (Participants) | 11 | 11 | 19 | 3
Ratio
  Day 1: number analyzed (Participants) | 0 | 11 | 0 | 0
  Day 1 |  | 0.9 [0.71 to 1.07] |  |
  Day 29 | 1.2 [0.89 to 1.68] | 4.3 [1.71 to 10.88] | 1.6 [0.49 to 5.48] | 1.0 [1.00 to 1.00]
  Day 57: number analyzed (Participants) | 10 | 10 | 0 | 0
  Day 57 | 1.1 [0.86 to 1.49] | 3.6 [1.42 to 9.33] |  |

6. Secondary Outcome: Number of ARCT-021-naïve Participants (Cohort 1a) With Seroconversion (Neutralizing Antibodies)
Description: Seroconversion was defined as a 4-fold increase in antibody titer/concentration from baseline. Data is presented for the number of participants seroconverting for neutralizing antibodies and immunoglobulin G (IgG) antibodies against the full-length SARS-CoV-2 recombinant spike protein antigen and spike protein receptor binding domain of the SARS-CoV-2 spike glycoprotein (RBD). ARCT-021-naïve participants were those participants whose first ARCT-021 vaccine administration occurred in this study (Cohort 1a). As pre-specified, data is presented for participants in Cohort 1a only.
Time Frame: Days 29, and 57
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a
Number analyzed (Participants) | 11
Participants
  Day 29 | 1
  Day 57: number analyzed (Participants) | 10
  Day 57 | 0

7. Secondary Outcome: Geometric Mean Concentration (GMC) of Serum SARS-CoV-2 Binding Antibodies
Description: GMC data are reported for the S (spike binding antibodies) analyte.
Time Frame: Cohorts 1a and 1b: Days 1, 29, 57, Cohort 2: Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary units per milliliter (AU/mL)
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2: Younger Adults | Cohort 2: Older Adults
Number analyzed (Participants) | 11 | 11 | 19 | 3
Arbitrary units per milliliter (AU/mL)
  Day 1: number analyzed (Participants) | 11 | 11 | 0 | 0
  Day 1 | 47.3 [24.06 to 93.12] | 310.6 [90.06 to 1071.18] |  |
  Day 29 | 1629.3 [770.41 to 3445.89] | 5319.8 [1817.81 to 15568.32] | 802.8 [349.23 to 1845.44] | 713.2 [178.25 to 2853.69]
  Day 57: number analyzed (Participants) | 10 | 10 | 0 | 0
  Day 57 | 1013.5 [501.13 to 2049.58] | 3088.1 [1172.00 to 8136.75] |  |

8. Secondary Outcome: GMFR in SARS-CoV-2 Binding Antibody Titers
Description: GMFR data are reported for the S (spike binding antibodies) analyte.
Time Frame: Cohort 1a: Days 29, 57, Cohort 1b: Days 1, 29, 57, and Cohort 2: Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2: Younger Adults | Cohort 2: Older Adults
Number analyzed (Participants) | 11 | 11 | 19 | 3
Ratio
  Day 1: number analyzed (Participants) | 0 | 11 | 0 | 0
  Day 1 |  | 7.2 [3.83 to 13.45] |  |
  Day 29 | 34.4 [16.76 to 70.69] | 136.5 [46.58 to 400.08] | 13.3 [3.94 to 44.75] | 29.6 [15.80 to 55.33]
  Day 57: number analyzed (Participants) | 10 | 10 | 0 | 0
  Day 57 | 20.4 [10.59 to 39.24] | 104.9 [34.62 to 317.74] |  |

9. Secondary Outcome: Number of ARCT-021-naïve Participants (Cohort 1a) With Seroconversion (Binding Antibodies)
Description: Seroconversion was defined as a 4-fold increase in antibody titer/concentration from baseline. Data is presented for the number of participants seroconverting for binding antibodies and immunoglobulin G (IgG) antibodies against the full-length SARS-CoV-2 recombinant spike protein antigen and spike protein receptor binding domain of the SARS-CoV-2 spike glycoprotein (RBD). ARCT-021-naïve participants were those participants whose first ARCT-021 vaccine administration occurred in this study (Cohort 1a). As pre-specified, data is presented for participants in Cohort 1a only.
Time Frame: Days 29, and 57
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a
Number analyzed (Participants) | 11
Participants
  Day 29 | 10
  Day 57: number analyzed (Participants) | 10
  Day 57 | 9

ADVERSE EVENTS:
Time Frame: Up to a maximum of approximately 12 months
Description: All-cause mortality is reported for all enrolled participants. Serious and other adverse events are reported in the Safety population for Cohort 1a, which included all participants who received Study vaccine in ARCT-021-02 only, and in the Longitudinal Safety population for Cohorts 1b and Cohort 2, which included all participants who received Study vaccine in ARCT- 021-01 and ARCT-021-02 (Cohort 1b) or ARCT-021-01 only (Cohort 2).
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2: Younger Adults | Cohort 2: Older Adults
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/25 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/25 | 0/16
Other Adverse Events (participants affected / at risk) | 3/12 | 1/12 | 3/25 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a (N=12) | Cohort 1b (N=12) | Cohort 2: Younger Adults (N=25) | Cohort 2: Older Adults (N=16)
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a (N=12) | Cohort 1b (N=12) | Cohort 2: Younger Adults (N=25) | Cohort 2: Older Adults (N=16)
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT04728347/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT04728347/SAP_002.pdf